CLINICAL TRIAL: NCT06949592
Title: Evaluation of Oral Bioavailability of the Phenolic Compounds in a Melissa Supplement: Double-blind, Randomized, Crossover Study
Brief Title: Oral Bioavailability of the Phenolic Compounds in a Melissa Supplement
Acronym: BIOLEMON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIOLEMON
Record Dates: First submitted 2025-04-18; First posted 2025-04-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): This arm receives 400 mg maltodextrin
  Interventions: Dietary Supplement: Placebo
- M_ML (Experimental): This arm receives 400 mg of M_ML. M_ML is a mixture of a polyphenol-rich Melissa officinalis extract, an acerola extract and vitamin B5.
  Interventions: Dietary Supplement: M_ML

INTERVENTIONS:
Dietary Supplement: Placebo — Intake of 400 mg placebo (maltodextrin; encapsulated) in the morning (09:00)
  Arms: Placebo
Dietary Supplement: M_ML — Intake of 400 mg M_ML (encapsulated) in the morning (09:00)
  Arms: M_ML
Dietary Supplement: M_ML — Intake of 400 mg M_ML (encapsulated) in the evening (19:00)
  Arms: M_ML

SUMMARY:
The objective of this study is to identify phenolic compound biomarkers of the intake of a mixture of Melissa officinalis extract, acerola extract and vitamin B5. This will be done through the study of their bioavailability and nutrikinetics by measuring their plasma concentrations and urinary excretion over 24h by means of high-performance liquid chromatography coupled with tandem mass spectrometry (HPLC-MS/MS). The study follows a cross-over, double-blind, randomized and placebo control design on 10 healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 60 years old.
* Agree to follow the dietary and exercise guidelines of the study.
* Sign the informed consent form.
* Be able to read, write, and speak Spanish and/or Catalan.

Exclusion Criteria:

* Body Mass Index (BMI) <18.5 kg/m² or ≥30 kg/m².
* Presence of intolerances or allergies related to polyphenols or any of the components of the products evaluated, such as acerola, maltodextrin, or Melissa officinalis.
* Use of medication that could affect the study results, including antibiotics, glucocorticoids, steroids, antidepressants (especially selective serotonin reuptake inhibitors (SSRIs), medications used to control sleep or stress, antipsychotics, anticonvulsants, oral contraceptives, beta-blockers, benzodiazepines, and antihypertensives.
* Regular consumption herbal or plant-based supplements. Participants who take multivitamin supplements may still participate in the study, provided they agree to stop taking them for 48 hours before and on the day of the intervention.
* Regular consumption of melatonin supplements. Participants who occasionally take melatonin may be included if they have had at least a one-week washout period since the last dose.
* Presence of disrupted sleep cycle or irregular sleep routines, such as shift workers (night or rotating shifts), or due to external factors such as recent or upcoming travel across time zones, or co-sleeping with a newborn/baby that disrupts sleep.
* Report self-perceived psychological stress, meaning they answer "yes" to the question: "Do you consider yourself to be severely stressed?"
* Self-reported trouble sleeping and/or falling asleep.
* To be diagnosed with anemia.
* Active smoker or have quit smoking less than 6 months ago.
* Consumption of alcoholic beverages: Men: 4 or more Standard Drink Units (SDUs)* daily or 28 SDUs weekly; Women: 2 or more SDUs daily or 17 SDUs weekly.
* Presence of liver, kidney, or gastrointestinal disease that may affect compound absorption and/or study results, such as: celiac disease, Crohn's disease, chronic kidney disease, active cancer in any digestive or renal organ, or hepatitis.
* Previous blood extraction and/or donation: ≥200 ml within 1 month prior to study inclusion, or ≥400 ml within 3 months prior to study inclusion.
* Have lost 3 kg or more in the past 3 months.
* Pregnant or planning to become pregnant.
* Currently breastfeeding.
* Unable to comply with the study protocol.
* Currently participating or have participated in a nutritional intervention study involving nutraceuticals or pharmaceuticals within the 30 days prior to inclusion in this study.
* Deemed unsuitable to participate in the study according to the judgment of the evaluator conducting the pre-selection.

One SDU is defined as the average alcohol content of a standard drink in terms of alcohol strength and volume. One SDU is approximately 10 grams of alcohol, which equals:1 glass of wine (120 ml), 1 beer (330 ml), 1 small liquor (25 ml); 2 SDUs equal: 1 glass of cognac or liqueur (55 ml),1 whisky (70 ml),1 mixed drink (75 ml).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Changes in plasma concentrations of phenolic metabolites after acute ingestion of the supplement/placebo | At baseline and at 0.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, and 24 hour after treatment intake.
  Plasma samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using liquid chromatography-time of light-mass spectometry (LC-qToF-MS). Results will be reported in nanomolar (nM).

SECONDARY OUTCOMES:
Change in plasma area under the curve (AUC) of phenolic metabolites after acute ingestion of the supplement/placebo | At baseline and at 0.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, and 24 hour after treatment intake.
  Plasma samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS.
Change in plasma maximal concentration (Cmax) of phenolic metabolites after acute ingestion of the supplement/placebo | At baseline and at 0.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, and 24 hour after treatment intake.
  Plasma samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS.
Change in plasma time to reach maximal concentration (Tmax) of phenolic metabolites after acute ingestion of the supplement/placebo | At baseline and at 0.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, and 24 hour after treatment intake.
  Plasma samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS.
Change in plasma half-life (T1/2) of phenolic metabolites after acute ingestion of the supplement/placebo | At baseline and at 0.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, and 24 hour after treatment intake.
  Plasma samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS.
Changes in 24h cumulative urinary excretion of phenolic metabolites after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in serum cortisol after acute ingestion of the supplement/placebo | At baseline and at 30.5 hour, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, and 24 hour after treatment intake.
  Serum samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using ECLIA (electrochemiluminescence immunoassay)
Changes in 24h cumulative urinary excretion of melatonin after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of 6-SMT (6-Sulfatoxymelatonin) after acute ingestion of the supplement/placebo | At baseline and at 3, 6, 10 and 24h after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of AFMK (N1-acetyl-N2-formyl-5-methoxykynuramine) after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of AMK (N1-acetyl-5-methoxykynuramine) after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of cortisol after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of cortisone after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of tetrahydrocortisol after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of allo-tetrahydrocortisol after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of 5-alfa-dihydrocortisol after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of 11-oxo-cortisol after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.
Changes in 24h cumulative urinary excretion of 11-oxo-corticosterone after acute ingestion of the supplement/placebo | At baseline and at 3 hour, 6 hour, 10 hour and 24 hour after treatment intake.
  Urine samples will be collected in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Concentrations will be analyzed using LC-qToF-MS, and transformed to total excretion through measured excreted urinary volume.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari Palou, PhD, Principal Investigator — Fundació Eurecat
Locations (1):
- Eurecat, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No